CLINICAL TRIAL: NCT05399238
Title: Thermography as a Non-ionizing Quantitative Tool for Diagnosing of Burning Mouth Syndrome
Brief Title: Thermography and Burning Mouth Syndrome
Acronym: TDSBA
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Director Oral Medicine, Universidad de Murcia
Other Study IDs: 3608/2021
Record Dates: First submitted 2022-05-17; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: The objective is to measure the temperature of the lingual dorsum
  Interventions: Device: The objective is to measure the temperature of the lingual dorsum
- Burning mouth syndrome: The objective is to measure the temperature of the lingual dorsum
  Interventions: Device: The objective is to measure the temperature of the lingual dorsum

INTERVENTIONS:
Device: The objective is to measure the temperature of the lingual dorsum — Subjects will make one visit to our clinic with burning mouth syndrome and control healthy . They will be asked to acclimate to room temperature for at least 20 minutes. Subjects are requested not to consume hot drinks or food for at least an hour before imaging and not to use any skin preparations.

SUMMARY:
Medical thermography is a noninvasive technique that allows an examiner to visualize and estimate the temperature of the body . This technique allows for an evaluation of the functionality of the structures, which is why it is considered a physiological test and records the variation in the surface temperature of the human body based on the infrared radiation emitted by the surface of that body .Subjects with burning mouth syndrome (BMS) have altered sensitivity and pain thresholds for thermal stimuli compared to a control group An objective of this study is to standardize temperature values derived from thermograms of the tongue in BMS .

DETAILED DESCRIPTION:
An objective of this study is to standardize temperature values derived from thermograms of the tongue in BMS

Subjects will make one visit to our clinic with burning mouth syndrome and control healthy . They will be asked to acclimate to room temperature for at least 20 minutes. Subjects are requested not to consume hot drinks or food for at least an hour before imaging and not to use any skin preparations. During the tests, infrared thermal images were taken immediately after subjects protruded their tongues forward and downward to the desired position

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed he patients were diagnosed with BMS according to the criteria of the International Classification of Headache Disorders

Exclusion Criteria:

* Fibromyalgia
* Fever
* Reflux
* Cancer,
* Oral infection,
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Burning mouth syndrome (BMS )patients and control healthy patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Measurement of temperature tongue | Day 1am . experimental subject and each control subject will be seen once for the administration of the thermography imagery
  Tongue temperature areas: tongue tip, middle, left lateral, right lateral,changes in colour pixels will be analysed to determine temperature changes since this is a measurement or diagnostic study using thermographic imagery, there is no health risk to the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

REFERENCES:
- [Background] Lv C, Wang X, Chen J, Yang N, Fisk I. A non-invasive measurement of tongue surface temperature. Food Res Int. 2019 Feb;116:499-507. doi: 10.1016/j.foodres.2018.08.066. Epub 2018 Aug 25. PMID 30716974
- [Background] Mo X, Zhang J, Fan Y, Svensson P, Wang K. Thermal and mechanical quantitative sensory testing in Chinese patients with burning mouth syndrome--a probable neuropathic pain condition? J Headache Pain. 2015;16:84. doi: 10.1186/s10194-015-0565-x. Epub 2015 Sep 24. PMID 26399417